CLINICAL TRIAL: NCT04145713
Title: Effects of Probiotic Mixture Supplementation and Evaluation of Intestinal Mucosal Tolerance and Gut Microbiome in Newborns With Perinatal Asphyxia Receiving Hypothermic Treatment: a Randomized, Multicentric, Blinded, Controlled Trial
Brief Title: Effects of Probiotic Mixture Supplementation and Evaluation of Intestinal Mucosal Tolerance and Gut Microbiome in Newborns With Perinatal Asphyxia Receiving Hypothermic Treatment
Acronym: VISNAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, Principal Investigator, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VISNAT
Record Dates: First submitted 2019-10-23; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Asphyxia Neonatorum; Morbidity;Newborn
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, blinded, multicentre
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: Probiotic mixture
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic mixture — The experimental intervention will consist in administrating a high-dose multi-strain probiotic (SIVOMIXXTM) for 30 days in addition to hypothermic therapy. The administration of probiotics will begin during the first 24 hours of hypothermia, at the dose of 1 capsule open in 5 millilitre of water. It will be administered daily for 30 days, either via nasogastric tube or orally.
  Arms: Probiotic group
Other: Placebo — The comparison intervention will consist in administrating placebo for 30 days in addition to hypothermic therapy. The administration of placebo will begin during the first 24 hours of hypothermia, at the dose of 1 capsule open in 5 millilitre of water. It will be administered daily for 30 days, either via nasogastric tube or orally.
  Arms: Placebo group

SUMMARY:
The VISNAT trial is a PILOT STUDY due to absence of previous evidences in literature on using probiotic in newborns with perinatal asphyxia.

It is designed as a randomized, placebo-controlled, blinded, multicentre superiority trial with two parallel groups and a primary outcome of mortality and/or disability at 18 months of age.

After informed consent is obtained from both parents, randomization will be performed as block randomization with a 1:1 allocation using a computer-generated allocation sequence, while the allocation concealment will be performed using locked bags.

Randomization data and allocation list will be stored in a secure place and will not be available to any of the components of the study apart of data collectors.

Participant files will be stored for a period of 10 years after completion of the study.

All the components of the study will be blinded including: participants and their parents, healthcare providers, outcome assessors, data collectors, data analysts.

ELIGIBILITY:
Inclusion Criteria:

* o Newborns with gestational age >/= 35 weeks and birth weight >/= 1800 grams

  o Intrapartum asphyxia defined according at least one of the following:
* APGAR index at 10 minutes </=5;
* Resuscitation with endotracheal tube or mask IPPV for more then 10 minutes;
* pH </= 7 or excess of base >/= 12 mmol/l on arterial blood gas (ABG) analysis within the first 60 minutes of life

  * Moderate/severe Hypoxic-ischemic encephalopathy assessed between 30 and 60 minutes of life according to Sarnat & Sarnat definition
  * Hypothermic treatment. According to the Italian national guidelines on Perinatal Asphyxia and Therapeutic Hypothermia, the hypothermic therapy will be started in the first six hours of life and will last 72 hours.

Exclusion Criteria:

* Inability to obtain the informed consent from both parents
* Congenital major malformations or syndromes o Surgical diseases

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 18 months
  Severe disability according to BAYLEY MENTAL DEVELOPMENT IINDEX
Mortality | 18 months
  Death

CONTACTS AND LOCATIONS:
Locations (1):
- Nicola Laforgia, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No